CLINICAL TRIAL: NCT05454371
Title: Investigation of Urinary Biomarkers for the Detection of Prostate Cancer
Acronym: URODETECT-WP2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is part of PhD trajectory and currently the trajectory is in the final phases without the official start of this recruitment.
Sponsor: Novosanis NV (Industry)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECO_CT29A
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer; Urine; Liquid Biopsy
Keywords: First-void urine; Liquid biopsy; Oncology; Biomarker; Colli-Pee
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample collection (Experimental): This is a prospective study in which urine samples will be collected from healthy volunteers and urine samples and a blood sample from cancer patients with breast- or prostate cancer. The participants will be asked to provide a urine sample collected with the ColliPee® device and fill out an online questionnaire to collect usability data.
  Interventions: Device: Colli-Pee UAS devices

INTERVENTIONS:
Device: Colli-Pee UAS devices — Colli-Pee UAS device variants will be evaluated during this study

SUMMARY:
The aim of this study is to investigate and possibly validate urinary biomarkers for prostate cancer. During this study the focus will be on aberrations of selected genes as prognostic or predictive value has been shown for these genes in tissue, CTC or blood derived cfDNA. Proteins will be explored in urine as well.

This is a prospective study in which urine samples will be collected from healthy volunteers and urine samples and a blood sample from cancer patients with prostate cancer. The participants will be asked to provide a urine sample collected with the ColliPee® device and fill out an online questionnaire to collect usability data. Thereafter, the urine sample will be aliquoted to be used in the study to investigate the different urinary analytes.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Being able to understand and read Dutch
* For cancer patients: being diagnosed with prostate cancer
* For healthy volunteers: being male

Exclusion Criteria:

* For cancer patients: suffering from a blood cancer
* For healthy volunteers: diagnosed with cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Detection (absence/presence) of specific urinary biomarker targets (AR-V7, TMPRSS2-ERG) for prostate cancer patients measured using ddPCR. | Through study completion, an average of 1 year.
  Comparison of target detection measured using ddPCR assays [positive, negative or copies/µL] in first-void urine samples from prostate cancer patients compared to age- and sex-matched healthy volunteers. (Proof of concept study)

SECONDARY OUTCOMES:
Detection (absence/presence) of specific biomarker targets (AR-V7, TMPRSS2-ERG) for prostate cancer patients measured using ddPCR. | Through study completion, an average of 1 year
  Comparison of target detection measured using ddPCR assays [positive, negative or copies/µL] in first-void urine samples from all study participants compared to blood testing using ddPCR. (Proof of concept study)
Usability characteristics of the Colli-Pee UAS devices. | Through study completion, an average of 1 year
  All study participants will receive a questionnaire regarding the usability characteristic of the Colli-Pee UAS devices. These questions cover physical information, previous experiences, and usability questions. When scores need to be given participants can score between 0 and 100%, in which 0% is a negative score and 100% is a positive score. When an opinion is asked participants can choose between very difficult, difficult, neutral, easy, and very easy. Analysis will be done using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No